CLINICAL TRIAL: NCT05081440
Title: A Multi-center, Prospective, Observational Study to Describe the siTuation of Blood Lipid mAnagement Among the Population With hypeRtension and/or Type 2 diabeTes in Community Health Center(START-CHC)
Brief Title: A Multi-center, Prospective, Observational Study to Describe the siTuation of Blood Lipid mAnagement Among the Population With hypeRtension and/or Type 2 diabeTes in Community Health Center
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Huashan Hospital (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Yong Li, PhD, MD, Huashan Hospital
Other Study IDs: START-CHC
Record Dates: First submitted 2021-10-05; First posted 2021-10-18 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Lipoprotein Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients diagnosed with hypertension or diabetes: Age ≥18 years; Patients with well-diagnosed hypertension (HTN) and/or type 2 diabetes (T2DM) and have been ill for ≥ 3 months; The patient underwent fasting lipid analysis in the past 1 month and the data was fully recorded

SUMMARY:
A multi-center, prospective, observational Study to describe the siTuation of blood lipid mAnagement among the population with hypeRtension and/or type 2 diabeTes in Community Health Center

ELIGIBILITY:
Inclusion Criteria:

1. The informed consent form (ICF) should be signed before conducting any research-related operations
2. Age ≥18 years
3. Patients with well-diagnosed hypertension (HTN) and/or type 2 diabetes (T2DM) and have been ill for ≥ 3 months
4. The patient underwent fasting lipid analysis in the past 1 month and the data was fully recorded

Exclusion Criteria:

1.Patients with well-diagnosed atherosclerotic cardiovascular disease (ASCVD) 2. Have received any form of lipid-lowering treatment within 4 weeks before the screening period 3. The patient is currently participating in any other clinical trial except this study

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 5000 patients with hypeRtension and/or type 2 diabeTes inCommunity Health Center
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
primary outcome | 2022.12.01
  To evaluate the blood lipid levels and current status of drug treatment in patients with CHC hypertension and/or type 2 diabetes Describe the characteristics of blood lipid treatment in patients with CHC with hypertension and/or type 2 diabetes with LDL-C between 2.6 and 4.1 mmol/L

SECONDARY OUTCOMES:
secondary outcome | 2022.12.01
  To evaluate the ASCVD risk stratification and the level of blood lipids in patients with CHC hypertension and/or type 2 diabetes.
  Evaluate the blood lipid level of patients with hypertension and/or type 2 diabetes in CHC with LDL-C between 2.6 and 4.1mmol/L (LDL-C/Non-HDL) To explore the compliance of patients with CHC hypertension and/or type 2 diabetes with LDL-C between 2.6 and 4.1 mmol/L for lipid-lowering therapy.